CLINICAL TRIAL: NCT05185414
Title: Combining Exome and Transcriptome Data to Unravel the Genetic Basis of the Lissencephalies
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Collaborators: Marguerite - Marie Delacroix Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: TRANSC_LIS
Record Dates: First submitted 2021-12-22; First posted 2022-01-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-11

CONDITIONS: Classical Lissencephalies and Subcortical Band Heterotopias
Keywords: Lissencephaly; rna sequencing
MeSH Terms: conditions — Classical Lissencephalies and Subcortical Band Heterotopias; Lissencephaly | interventions — Phlebotomy

STUDY DESIGN:
Intervention Model Description: Diagnostic track: apply rna sequencing on lissencephaly patients without genetic diagnosis to establish diagnosis
  Research track: apply rna sequencing on lissencephaly patient with an established genetic diagnosis to investigate additional diagnositc yield, suited sampling tissue and rna patterns
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RNA sequencing in genetically solved lissencephaly cases (Other): RNA expression patterns in lissencephalies. RNA sequencing will be applied to the genetically solved lissencephaly cases. The acquired information on RNA expression patterns will be implemented in unsolved lissencephaly cases.
  Interventions: Diagnostic Test: Venipuncture and skin biopsy for RNA extraction
- RNA sequencing in genetically unsolved lissencephaly cases (Other): Obtain a genetic diagnosis in unsolved lissencephaly cases by implementation of RNA expression patterns obtained in arm 1.
  Interventions: Diagnostic Test: Venipuncture and skin biopsy for RNA extraction

INTERVENTIONS:
Diagnostic Test: Venipuncture and skin biopsy for RNA extraction — * Blood sampling (standard venipuncture)
  * Skin biopsy (fibroblasts)

SUMMARY:
Malformations of cortical development (MCD) are a heterogenous group of brain malformations including lissencephaly, heterotopia and polymicrogyria. The lissencephaly spectrum (including lissencephaly, pachygyria and subcortical band heterotopia) is a well-defined group of MCD with a strong monogenetic basis. Using current molecular techniques, a causative variant is detected in approximately 80% of individuals with lissencephaly. In a routine diagnostic setting, exome-based gene panels are most frequently used while whole exome sequencing (WES) and whole genome sequencing (WGS) are increasingly being implemented. Both techniques have their shortcomings including the detection of small copy number variants, the identification of pathogenic variants in non-coding regions as well as variant interpretation. The parallel use of quantitative RNA sequencing, measuring differences in RNA expression could be a possible solution for these shortcomings. The proposed research project will for the first time 1) evaluate the added value of WES/WGS combined with quantitative RNA sequencing for the identification of novel genes in individuals with lissencephaly, 2) identify the optimal sampling tissue for RNA sequencing in complex neurological phenotypes and 3) use RNA expression data to provide an evidence base for the current lissencephaly classification.

DETAILED DESCRIPTION:
As mentioned before, lissencephalies have a strong monogenetic base in contrast to other brain malformations. Approximately 80% percent of the lissencephalies can be genetically diagnosed by standard WES or WGS.1 In the remaining 20% percent of unsolved cases quantitative RNA sequencing could make a considerable difference. By identifying RNA expression patterns in lissencephalies we will try to provide unsolved lissencephaly cases with a genetic diagnosis. A genetic diagnosis is im-portant in terms of predicting associated problems, follow-up, prognosis and in some cases family planning (e.g. pre-implantation genetic testing). This study will also investigate the additional diagnostic yield of RNA sequencing in lissencephalies and by extension in the MCD spectrum. And, if indicated, the feasibility of implementing RNA sequencing in the standard diagnostic work-up.

High efficiency in identifying new pathogenic variants and novel gene annotation can be expected because of the strong monogenetic base. These novel variants and gene annotation are indispensable for better understanding the origin and pathophysiology of the lissencephaly spectrum and neuronal migration.

The functional impact of newly discovered genes can be further investigated by the innovative CRISPR-Cas9 method. This gene-editing technique allows researchers to create knock-out or even knock-in genes, as an opportunity to investigate novel annotated genes and their functional consequences. Although it is beyond the scope of this study, it is an interesting item for future joined research projects, within our research group or in collaboration with others. During this study, also genetically diagnosed lissencephaly cases will be subjected to RNA sequencing. The current classifi-cation of lissencephalies is based on pathogenic variants and biological pathways. Alterations in RNA-expression pattern could possibly shine a new light on this classification.

This study will also evaluate which sampling tissues are most suited for RNA extraction and sequencing. Considerations to make include the targeted quality of the extracted RNA and differences in tissue-specific gene expression. Mouth swaps, although non-invasive, are not suited for RNA extraction because of the natural oral flora with multiple viruses and bacteria (exogenous genetic material). Fibroblast-derived RNA is considered to be of good quality, but a skin biopsy is required and considered relatively invasive. Whole blood is obtained by minimal invasive techniques, but gene expression may be of poorer quality compared to fibroblasts.

The first part of the study is performed in a diagnostic setting in unsolved lissencephaly cases. Fibroblasts will be obtained by skin biopsy (punch). RNA seq data will be extracted from fibroblasts and blood. This RNA seq data will be analyzed in search for new pathogenic variants. When new pathogenic variants are identified in the RNA seq data, existing WES data will be reanalyzed. If neces-sary, subsequent WGS will be performed. When a genetic diagnosis is obtained, RNA seq and WES/WGS data will be transferred to the research part of the study.

A second part of the study is performed in a research setting. Lissencephaly patients with a genetic diagnosis will be proposed to donate a skin biopsy and . RNA seq data will be extracted from fibroblasts and blood as in the diagnostic track. In the RNA seq data two items will be observed. Firstly, has RNA seq data extracted from fibroblasts a major advantage over RNA seq data extracted from blood in terms of variant detection? Secondly, can RNA patterns be identified in common affected pathways?

ELIGIBILITY:
Inclusion Criteria:

Overall:

* anomaly on MRI of the lissencephaly spectrum (lissencephaly, pachygyria, subcortical band heterotopia

Diagnostic track:

* No established genetic diagnosis by conventional WES/WGS

Research track:

* An established genetic diagnosis by conventinal WES/WGS

Exclusion Criteria:

* No anomaly of the lissencephaly spectrum on MRI

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-01 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Additional diagnostic yield of RNA seq in clinical practice | 4 years
  Does combined WES/WGS and rna seq approach increase the diagnostic yield for lissencephalies compared to conventional WES/WGS? If yes, to what extend? Can it be implemented in the standard diagnostic flowcharts?
  This study will combine WES and (quantitative) RNA sequencing in a subgroup of the MCD spectrum. It is estimated that 80% percent of the lissencephalies can be genetically diagnosed by standard WES or WGS, leaving +/- 20% of cases unsolved. WGS will be applied in specific cases where WES remains negative (e.g. alterations in RNA expression pattern). This approach has never been applied to MCD before. Most accurate numbers can be derived from the few case series that have been published, where quantitative RNA sequencing was found to extend the diagnostic yield between 7 and 35%. These results are based on small case series, consisting of heterogenous phenotypes and are difficult to extrapolate to the proposed research set-up based on a well-delineated phenotype.

SECONDARY OUTCOMES:
Suited sampling tissue for rna sequencing | 4 years
  What is the added value of fibroblasts sampling compared to standard blood sampling for quantitative RNA sequencing in the context of lissencephalies?
  Literature suggests that gene expression fluctuates between different tissues. Small case series suggest that the expression of genes involved in neurological phenotypes is better in fibroblast tissue compared to whole blood. In three out of six cases the pathogenic variant was not discovered by RNA analysis on whole blood, nevertheless that RNA analysis on fibroblast tissue was able to uncover all six pathogenic variants (Murdock et al. 2020). An objective of this study is to compare results of quantitative RNA sequencing on whole blood versus fibroblasts in a large case series. Pros and cons of blood sampling versus fibroblasts have to be taken into account.
rna expression in lissencephalies | 4 Years
  The number of genes involved in the lissencephaly spectrum remains limited. Besides identify-ing new genes involved in lissencephaly, a third study objective will focus on the RNA expression pattern in known lissencephaly genes. A total of 21 lissencephaly genes have been described (Di Donato et al. (2018)) and others including 11 genes in which alterations are seen more frequently. By performing RNA sequencing on blood and fibroblast samples from patients with known pathogenic variants in these genes, we will try to identify RNA sequencing patterns and, if possible, biomarkers specific for these genes or groups of genes. This will enable us to 1) to predict the genes or pathways to focus on in patients with undiagnosed lissencephalies and 2) to better understand phenotype / genotype correlations and possibly 3) to make an alternative classification of lissencephalies.

CONTACTS AND LOCATIONS:
Overall Officials: Ellen RIJCKMANS, Dr, Principal Investigator — UZ Brussel - Vrije Universiteit Brussel
Locations (1):
- UZ Brussel, Jette, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: No
Might change in the future

REFERENCES:
- [Background] Di Donato N, Timms AE, Aldinger KA, Mirzaa GM, Bennett JT, Collins S, Olds C, Mei D, Chiari S, Carvill G, Myers CT, Riviere JB, Zaki MS; University of Washington Center for Mendelian Genomics; Gleeson JG, Rump A, Conti V, Parrini E, Ross ME, Ledbetter DH, Guerrini R, Dobyns WB. Analysis of 17 genes detects mutations in 81% of 811 patients with lissencephaly. Genet Med. 2018 Nov;20(11):1354-1364. doi: 10.1038/gim.2018.8. Epub 2018 Apr 19. PMID 29671837
- [Background] Gonorazky HD, Naumenko S, Ramani AK, Nelakuditi V, Mashouri P, Wang P, Kao D, Ohri K, Viththiyapaskaran S, Tarnopolsky MA, Mathews KD, Moore SA, Osorio AN, Villanova D, Kemaladewi DU, Cohn RD, Brudno M, Dowling JJ. Expanding the Boundaries of RNA Sequencing as a Diagnostic Tool for Rare Mendelian Disease. Am J Hum Genet. 2019 Mar 7;104(3):466-483. doi: 10.1016/j.ajhg.2019.01.012. Epub 2019 Feb 28. PMID 30827497
- [Background] Severino M, Geraldo AF, Utz N, Tortora D, Pogledic I, Klonowski W, Triulzi F, Arrigoni F, Mankad K, Leventer RJ, Mancini GMS, Barkovich JA, Lequin MH, Rossi A. Definitions and classification of malformations of cortical development: practical guidelines. Brain. 2020 Oct 1;143(10):2874-2894. doi: 10.1093/brain/awaa174. PMID 32779696
- [Background] Murdock DR, Dai H, Burrage LC, Rosenfeld JA, Ketkar S, Muller MF, Yepez VA, Gagneur J, Liu P, Chen S, Jain M, Zapata G, Bacino CA, Chao HT, Moretti P, Craigen WJ, Hanchard NA; Undiagnosed Diseases Network; Lee B. Transcriptome-directed analysis for Mendelian disease diagnosis overcomes limitations of conventional genomic testing. J Clin Invest. 2021 Jan 4;131(1):e141500. doi: 10.1172/JCI141500. PMID 33001864